CLINICAL TRIAL: NCT05102292
Title: An Open Label, Multicenter Phase Ib/II Clinical Study to Evaluate Efficacy , Safety and PK of HLX208 in Advanced Anaplastic Thyroid Cancer (ATC) With BRAF V600 Mutation
Brief Title: The Efficacy and Safety of HLX208 in Advanced Anaplastic Thyroid Cancer (ATC) With BRAF V600 Mutation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-ATC201
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Anaplastic Thyroid Cancer; ATC
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — CCT239065

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX208 (Experimental): Participants receive HLX208 450mg bid po
  Interventions: Drug: HLX208

INTERVENTIONS:
Drug: HLX208 — HLX208 450mg bid po
  Other Names: BRAF V600E inhibitor

SUMMARY:
The purpose of this study was to assess efficacy, safety and PK in anaplastic thyroid cancer (ATC) given HLX208 (BRAF V600E inhibitor).

ELIGIBILITY:
Inclusion Criteria:

1. Age>=18Y;
2. Good Organ Function;
3. Expected survival time ≥ 3 months;
4. Advanced BRAF V600 ATC that have been diagnosed histologically;
5. At least one measurable lesion as per RECIST v1.1;
6. ECOG score 0-1.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Previous treatment with BRAF inhibitors or MEK inhibitors;
3. A history of other malignancies within two years, except for cured cervical carcinoma in situ, basal cell carcinoma of the skin;
4. Severe active infections requiring systemic anti-infective therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate(assessed by independent radiological review committee (IRRC) based on the RECIST Version 1.1)

SECONDARY OUTCOMES:
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (PFS) (assessed by IRRC and the investigator as per RECIST v1.1 )
OS | from the date of first dose until the date of death from any cause，assessed up to 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Affiliated Oncology Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No